CLINICAL TRIAL: NCT02655588
Title: A Computerized Intervention for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Stone (Other)
Collaborators: Harvard University (Other)
Responsible Party: Sponsor-Investigator, William Stone, Assistant Professor, Beth Israel Deaconess Medical Center
Organization: Beth Israel Deaconess Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P000384
Record Dates: First submitted 2016-01-05; First posted 2016-01-14 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ImbPST (Experimental): ImbPST Arm: Participants in this arm will interact with imbPST program which provides a simulated therapy session based on the Problem Solving Treatment-Primary Care (PST-PC) treatment manual used in depression clinical trials . imbPST via a "virtual" therapist (presented via audio and video) provides programmed instructions on the steps and skills of problem solving, emotional support, and tailored feedback to the user's input.
  Interventions: Behavioral: Interactive Media-Based Problems Solving Treatment
- Control Group (No Intervention): Control Arm: Participants in this group will not receive any treatment for their depression and their depressive symptoms will be monitored for 6 to 9 weeks

INTERVENTIONS:
Behavioral: Interactive Media-Based Problems Solving Treatment
  Arms: ImbPST

SUMMARY:
The primary purpose of this study is to examine how much change in depressive symptoms will be observed in persons who use an electronic Problem Solving Treatment (imbPST) compared to a control group at pre-, mid-point, and post-test assessments.

DETAILED DESCRIPTION:
An interactive multimedia computer-based treatment program was developed to provide an electronic version of problem solving therapy for depression (imbPST). The program was entirely automated and did not require the involvement of a live clinician, even though it was designed to provide a "virtual therapy" experience that feels more like interacting with a person than with a computer. The imbPST program was built to help individuals who did not have access to traditional therapy due the living conditions or individual preferences (e.g. rural, poor and persons desiring privacy or with significant time constraints). This computer-based treatment of depression offered several advantages. It can be used anywhere without a therapist present, and offered a standardized and consistent therapeutic approach.

The aim of this study is to reduce symptoms of depression in subjects through the use of a new, electronic Problem Solving Treatment (imbPST). Adult participants with moderate to severe depression symptoms are randomly assigned to either treatment or a wait-list condition. The Beck Depression Inventory-II was used as the primary outcome measure

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older.
2. Present symptoms from the following criteria based on the Diagnostic & Statistical Manual of Mental Disorders-IV-Text Revision (DSM-IV-TR): Major Depressive Episode, Mood Disorder Due to a General Medical Condition and/or Adjustment Disorder with Depressed Mood.
3. Depression must be the primary diagnosis and not occur secondary to any another diagnosis such as Post-Traumatic Stress Disorder (PTSD), social phobia, or complicated bereavement, though comorbid diagnoses (e.g., anxiety disorders and PTSD) will not be exclusionary unless they are primary, except as specified below.
4. Not receiving psychological treatment (e.g., face to face) at the time of the study.
5. Not currently be receiving Problem Solving Treatment in any other context.
6. Not reporting/reported suicidal attempts in the year prior to their participation in the study.
7. Be able to write and speak English according to Rapid Estimate of Adult Literacy in Medicine (REALM test scores)

Exclusion Criteria:

1. Current suicidal ideation, history of suicidal attempts or self-injurious behavior at any point during the protocol.
2. Have been diagnosed with schizophrenia, bipolar I disorder, with psychosis, other disorder with psychotic symptoms, and/or brain injuries that includes loss of consciousness > 15 minutes and / post-traumatic amnesia of any duration.
3. Any history of treatment with anti-psychotic medication.
4. A felony conviction.
5. Any current or recent (i.e. within the previous 6 months) substance abuse/dependence diagnosis (other than nicotine or caffeine).
6. Current psychological treatment (e.g., face to face).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-09; Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Symptoms of Depression will be assessed by using the Beck Depression Inventory II | Within the first 9 weeks after initiating treatment.
  Self-report measure for symptoms of depression

SECONDARY OUTCOMES:
Software usability will be measured by the System Usability Scale | at baseline (week 0),and post-treatment ( week 9)
  Self-report measure
Symptoms of Depression will be assessed by using the Hopkins Symptom Checklist 20-item Depression Scale ( Self-report) | Within the first 9 weeks after initiating treatment.
  Self-report measure for symptoms of depression

CONTACTS AND LOCATIONS:
Overall Officials: William Stone, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnau RC, Meagher MW, Norris MP, Bramson R. Psychometric evaluation of the Beck Depression Inventory-II with primary care medical patients. Health Psychol. 2001 Mar;20(2):112-9. doi: 10.1037//0278-6133.20.2.112. PMID 11315728
- [Background] Hegel, M.T., & Arean, P.A. (2003) Problem-solving Treatment for Primary Care (PST-PC): A Treatment Manual for Depression
- [Background] Munoz RF, Cuijpers P, Smit F, Barrera AZ, Leykin Y. Prevention of major depression. Annu Rev Clin Psychol. 2010;6:181-212. doi: 10.1146/annurev-clinpsy-033109-132040. PMID 20192789
- [Background] Proudfoot J, Goldberg D, Mann A, Everitt B, Marks I, Gray JA. Computerized, interactive, multimedia cognitive-behavioural program for anxiety and depression in general practice. Psychol Med. 2003 Feb;33(2):217-27. doi: 10.1017/s0033291702007225. PMID 12622301
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Heinzelmann PJ, Lugn NE, Kvedar JC. Telemedicine in the future. J Telemed Telecare. 2005;11(8):384-90. doi: 10.1177/1357633X0501100802. PMID 16356311
- [Background] Beck, A.T., Steer, R.A., & Garbin, M.C. (1988).Psychometric properties of the Beck Depression Inventory: Twenty-five years of evaluation. Clinical Psychology Review
- [Background] Lipman RS, Covi L, Shapiro AK. The Hopkins Symptom Checklist (HSCL)--factors derived from the HSCL-90. J Affect Disord. 1979 Mar;1(1):9-24. doi: 10.1016/0165-0327(79)90021-1. PMID 162184
- [Background] Thornett AM, Mynors-Wallis LM. Credibility of problem-solving therapy and medication for the treatment of depression among primary care patients. Med Sci Monit. 2002 Mar;8(3):CR193-6. PMID 11887035